CLINICAL TRIAL: NCT04048668
Title: Transcranial Direct Current Stimulation to Enhance Language Recovery in Patients With Aphasia After Subacute Stroke
Brief Title: tDCS to Treat Subacute Aphasia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Suspended due to COVID-19
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 813736
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Aphasia; Stroke, Acute
Keywords: non-invasive brain stimulation; tDCS
MeSH Terms: conditions — Aphasia; Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tDCS (Active Comparator): 2mA for 20 minutes
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS (Sham Comparator): 30 second ramp-up / ramp-down for 20 minutes
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — tDCS is a non-invasive brain stimulation technique by which very small electrical currents (2 mA) are applied to the scalp.
  Other Names: Standard of Care Speech Therapy

SUMMARY:
This study proposes to use transcranial direct current stimulation (tDCS), a technique by which a very small electrical current (2 mA) is applied to the scalp, along side speech therapy in patients with subacute stroke and aphasia in order to enhance language recovery. Aphasic patients in an inpatient neurorehabilitation facility who have experienced a stroke between one week and three months prior to enrollment will be invited to participate. Participants will receive either real or sham tDCS to the left hemisphere of the brain for a minimum of 5 consecutive sessions to up-to a max of 10 sessions depending on the length of their rehab stay . Stimulation will be paired with with the patient's normal speech therapy schedule. Participant's language skills will be assessed at baseline and immediately after the last session of therapy in order to determine whether tDCS is associated with either transient or persistent improvement in language.

DETAILED DESCRIPTION:
Speech therapy is the standard of care nationwide in treating individuals who have had a stroke and are now experiencing aphasia. Speech therapy can help to rehabilitate language skills and supplement function by teaching alternate strategies for communication; however, these benefits often leave room for further improvement. Researchers have focused their efforts in combining speech therapy with other techniques to boost the effects. In this study, we will combine speech therapy with non-invasive brain stimulation, specifically transcranial direct current stimulation (tDCS), in the hopes of significantly improve language in subacute aphasia patients.

This is a double-blind, randomized, sham-controlled pilot project, where inpatients with subacute stroke and aphasia will be recruited from the Penn Institute for Rehabilitation Medicine hospital (PIRM). The typical patient admitted to PIRM is approximately 1-2 weeks post-stroke. Upon enrollment, baseline aphasia severity will be characterized using standardized measures such as the Western Aphasia Battery (WAB), Pyramids and Palm Trees (PPT) and Philadelphia Naming Test (PNT) by the patient's speech therapist. Subjects will subsequently be randomized to undergo either real or sham tDCS. Subjects will then undergo a minimum of 5-consectuive stimulation session (Monday-Friday) and maximum of 10-consecutive stimulation sessions (Monday-Friday) of either real or sham tDCS. During stimulation, subjects will receive either real tDCS at a current of 2.0 mA for 20 minutes or sham stimulation for an equivalent period of time with a 30sec ramp-up/ramp-down. Sham stimulation mimics real stimulation closely; most subjects cannot distinguish between real and sham tDCS. During stimulation visits subjects will concurrently participate in their regular speech therapy treatment. Speech Therapy will be administered by their speech therapist and will follow whatever protocol the therapist deems useful for standard of care treatment of their aphasia. An immediate follow-up session will also take place, subjects will repeat language batteries including the WAB, PPT and PNT.

ELIGIBILITY:
Inclusion Criteria:

* 1. Presence of aphasia attributable to stroke that occurred between 7 days and 3 months (inclusive) prior to inclusion in the study.
* 2. Must be able to understand the nature of the study, and give informed consent.
* 3. English must be their native language where "native" is defined as learning English before the age of 6

Exclusion Criteria:

* 1. History of chronic, serious, or unstable neurologic illness(es) other than stroke
* 2. Current unstable medical illness(es)
* 3. History of reoccurring seizures or epilepsy
* 4. Current abuse of alcohol or drugs
* 5. Active or History of major psychiatric disorder
* 6. Pregnancy
* 7. Subjects with metallic objects in the face or head other than dental apparatus such as braces, fillings, and implants.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Aphasia Severity | Baseline, Immediate Follow-up
  Measured by WAB AQ score. A higher score indicated better language function. Scores can range from 0-100 with any score over 93 considered "recovered".

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Institute for Rehabilitation Medicine, Philadelphia, Pennsylvania, United States